CLINICAL TRIAL: NCT05165264
Title: A National, Prospective, Non-interventional Study (NIS) of Nivolumab Plus Chemotherapy in First Line Treatment of Adult Patients With HER2 Negative Advanced or Metastatic Gastric, Gastro-oesophageal Junction or Oesophageal Adenocarcinoma Whose Tumours Express PD-L1 With a CPS ≥5
Brief Title: A Study of Nivolumab Plus Chemotherapy in First Line Treatment of Adult Participants With Advanced or Metastatic Gastric Cancer
Acronym: INGA
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8EC
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
Keywords: OPDIVO®; Nivolumab; Advanced or Metastatic; Gastric Cancer; Prospective Study; Gastro-oesophageal junction; Oesophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with previously untreated advanced or metastatic gastric cancer (GC), gastro-oesophageal junction (GEJ) or oesophageal adenocarcinoma (EAC)

SUMMARY:
The purpose of this observational study is to assess the effectiveness and safety of nivolumab in participants with previously untreated advanced or metastatic Gastric Cancer (GC), Gastro-oesophageal Junction (GEJ) Adenocarcinoma, or Oesophageal Adenocarcinoma (EAC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HER2 negative advanced or metastatic HER2-negative GC, GEJ adenocarcinoma or EAC whose tumours express PD-L1 with a CPS ≥ 5
* Whose physician has decided to start a treatment with nivolumab (according to the German marketing authorization) for the treatment of GC, GEJ adenocarcinoma or EAC and prior to study participation

Exclusion Criteria:

* Previous malignancy within 3 years or concomitant malignancy, except: those with a 5-year overall survival rate of more than 90%, e.g. non-melanomatous skin cancer or adequately treated in situ cervical cancer.
* Participants currently included in an interventional clinical trial for their advanced or metastatic GC, GEJ adenocarcinoma or EAC. Participants who have completed their participation in an interventional trial or who are not receiving any study drug anymore and who are only in the follow-up Phase for OS can be enrolled. For blinded studies, the study drug administered needs to be known at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include participants with previously untreated advanced or metastatic GC, GEJ adenocarcinoma or EAC that will be enrolled continuously.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months
  Defined as time since initial diagnosis and treatment with nivolumab to either the first disease progression date or last known tumour assessment date, or death due to any cause, whichever occurs first.
Overall response rate (ORR) | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months
  Defined as investigator assessed complete response, partial response, stable disease, or progressive disease.
Duration of response | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months
  Defined as time from response to progression
Incidence of Adverse Events (AEs) | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months
Overall Survival (OS) | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months
  Defined as time since initial diagnosis and treatment with nivolumab until date of death due to any cause.
OS measured by Programmed Death-Ligand 1 (PD-L1) combined positive score (CPS) | From initial diagnosis and treatment with nivolumab until date of death due to any cause, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Hamburg, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html